CLINICAL TRIAL: NCT00005016
Title: The Experiences and Needs of Parents Continuing a Pregnancy Following Abnormal Prenatal Results: The Case of Holoprosencephaly
Brief Title: Study of the Experiences and Needs of Parents Continuing a Pregnancy Following a Prenatal Diagnosis of Holopresencephaly
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 000104; 00-HG-0104
Record Dates: First submitted 2000-04-04; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-03

CONDITIONS: Holoprosencephaly
Keywords: Fetal Anomaly; Genetic Counseling; Prenatal Diagnosis; Psychosocial Issues; Qualitative; HPE; Holoprosencephaly
MeSH Terms: conditions — Holoprosencephaly; Congenital Abnormalities

SUMMARY:
This study will examine the experiences of parents who decided to continue a pregnancy after receiving a prenatal diagnosis of holopresencephaly (HPE). HPE results from a genetic defect that can cause facial abnormalities such as cleft lip and cleft palate, learning disabilities, muscle weakness, problems with digestion, sleep and muscle control, and other disabilities. The severity of symptoms varies greatly among affected children.

Parents whose child was diagnosed before birth with HPE may be eligible for this study. It involves a one-time interview that takes from about 45 to 60 minutes. The interview is conducted either in person or by telephone and consists of three parts, as follows:

1. The experience of receiving the diagnosis of HPE during the pregnancy < includes general questions such as when and how HPE was diagnosed, what kind of information the parent received, the parent's reaction to the diagnosis, what genetic counseling, if any, the parents received, and so forth.
2. Emotional and informational needs < includes questions about the parent's specific emotional and informational needs from the time of diagnosis until the baby's birth, and the parent's reactions to support that was given.
3. Questionnaire < includes questions about the parent and his or her child, such as the parent's age, gender, marital status, and religious background, the child's age, gender, medical problems, and so forth. The questionnaire will be completed verbally for telephone interviews and in writing for in-person interviews. The interview will be tape-recorded and will be kept confidential.

Information from this study will provide health professionals, including genetic counselors, more effective strategies for helping other parents who face similar prenatal diagnoses.

DETAILED DESCRIPTION:
Holoprosencephaly (HPE) is a condition that when found prenatally offers parents a poor but often uncertain prognosis for their baby. Parents that continue the pregnancy given this diagnosis are left to endure the remainder of the pregnancy and the ambiguity involved in this highly variable condition. Previous studies have examined the psychological and social impact of prenatal diagnosis on parents and the outcomes of the pregnancy in conditions such as Down syndrome and sex chromosome abnormalities. Because the majority of parents receiving abnormal prenatal information terminate their pregnancies, most studies have focused on these parents' experiences, specifically the mothers'. However, little is known about the experiences of parents (both fathers and mothers) continuing a pregnancy given abnormal prenatal information especially in highly variable conditions such as HPE.

In this study, the experiences and needs of parents who received the diagnosis of HPE prenatally will be explored. Study participants will be drawn from several sites that include an existing molecular diagnostic protocol for HPE at the University of Pennsylvania, clinical patients seen at the University of Michigan, HPE family resources, and an upcoming conference on HPE to be held in April of 2000. Through semi-structured interviews, fathers and mothers of children with HPE who were diagnosed prenatally will be asked to talk individually about their experiences of receiving the diagnosis and continuing with the pregnancy. Their perceived informational, emotional and supportive needs at that time will be explored. In addition, their thoughts on the health care professionals' role in meeting these needs will be discussed. A brief questionnaire following the interview will gather quantitative data to serve as descriptors of the population and to help interpret the qualitative findings. The questionnaire includes demographic questions as well as a scale measuring tolerance for ambiguity and questions regarding the parent's perceived severity of their child's diagnosis of HPE.

Interviews will be analyzed qualitatively through thematic analysis. Specifically, recurring themes that emerge from interview transcripts will be analyzed for content and patterns. In addition, descriptive statistics will be applied to the questionnaire data and will be used to aid in the interpretation of the qualitative findings. An exploration of the experiences and needs of fathers and mothers who receive the diagnosis of HPE prenatally will offer a better understanding for health care professionals, specifically genetic counselors, regarding their role in working with parents continuing a pregnancy given prenatal information about a fetal anomaly.

ELIGIBILITY:
Parents, both fathers and mothers, of a child with HPE if they received their child's diagnosis of HPE prenatally either through ultrasound or prenatal testing such as CVS or amniocentesis.

Must have continued pregnancy after HPE diagnosis.

Must be over the age of 18.

Will not be excluded on the basis of single-parent status or of refusal of one parent to participate.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 2000-03; Study Completion 2001-02

CONTACTS AND LOCATIONS:
Locations (1):
- National Human Genome Research Institute (NHGRI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Beeson D, Golbus MS. Decision making: whether or not to have prenatal diagnosis and abortion for X-linked conditions. Am J Med Genet. 1985 Jan;20(1):107-14. doi: 10.1002/ajmg.1320200113. No abstract available. PMID 3970063
- [Background] Chitty LS, Barnes CA, Berry C. Continuing with pregnancy after a diagnosis of lethal abnormality: experience of five couples and recommendations for management. BMJ. 1996 Aug 24;313(7055):478-80. doi: 10.1136/bmj.313.7055.478. No abstract available. PMID 8776321
- [Background] Drugan A, Greb A, Johnson MP, Krivchenia EL, Uhlmann WR, Moghissi KS, Evans MI. Determinants of parental decisions to abort for chromosome abnormalities. Prenat Diagn. 1990 Aug;10(8):483-90. doi: 10.1002/pd.1970100802. PMID 2267225